CLINICAL TRIAL: NCT04632992
Title: MyTACTIC: An Open-Label Phase II Study Evaluating Targeted Therapies in Patients Who Have Advanced Solid Tumors With Genomic Alterations or Protein Expression Patterns Predictive of Response
Brief Title: A Study Evaluating Targeted Therapies in Participants Who Have Advanced Solid Tumors With Genomic Alterations or Protein Expression Patterns Predictive of Response
Acronym: MyTACTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML42439
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Advanced Unresectable or Metastatic Solid Malignancy
MeSH Terms: interventions — entrectinib; inavolisib; alectinib; ipatasertib; atezolizumab; Ado-Trastuzumab Emtansine; pertuzumab; Trastuzumab; tucatinib; Paclitaxel; Tiragolumab; pralsetinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Arm A: Entrectinib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for ROS1 gene fusion.
  Interventions: Drug: Entrectinib
- Arm B: Inavolisib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for PI3KCA activating mutation.
  Interventions: Drug: Inavolisib
- Arm C: Alectinib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for ALK rearrangement tumors.
  Interventions: Drug: Alectinib
- Arm D: Ipatasertib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for either AKT1/2/3 activating mutation or PTEN loss/loss of function.
  Interventions: Drug: Ipatasertib
- Arm E: Atezolizumab + Investigator's Choice of Chemotherapy (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for either tumor mutational burden (TMB) high or microsatellite instability (MSI) high/deficient mismatch repair (dMMR).
  Interventions: Drug: Atezolizumab; Drug: Investigator's Choice of Chemotherapy
- Arm F: Trastuzumab Emtansine + Atezolizumab (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for human epidermal growth factor receptor 2 (HER2) mutations or amplification without known TMB high or MSI high/dMMR.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab Emtansine
- Arm G: PH FDC SC (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for HER2 mutation or amplification without known TMB high or MSI high/dMMR.
  Interventions: Drug: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf
- Arm H: PH FDC SC + Investigator's Choice of Chemotherapy (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for HER2 mutation or amplification without known TMB high or MSI high/dMMR.
  Interventions: Drug: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Drug: Investigator's Choice of Chemotherapy
- Arm I: Trastuzumab Emtansine + Tucatinib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for HER2 mutation or amplification without known TMB high or MSI high/dMMR.
  Interventions: Drug: Trastuzumab Emtansine; Drug: Tucatinib
- Arm J: Trastuzumab Emtansine + Atezolizumab (Experimental): Participants in this treatment arm must have positive tumor biomarker results for HER2 mutation or amplification and TMB high or MSI high/dMMR.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab Emtansine
- Arm K: Ipatasertib + Atezolizumab (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for PI3KCA activating mutation.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab
- Arm L: Ipatasertib + Atezolizumab (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for either AKT1/2/3 activating mutation or PTEN loss/loss of function.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab
- Arm M: Ipatasertib + Paclitaxel (Experimental): Participants in this treatment arm must have a positive tumor biomarker results for PI3KCA activating mutations and either AKT1/2/3 activating mutation or PTEN loss/loss of function.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Arm N: Atezolizumab + Tiragolumab (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for either TMB high or MSI high/dMMR.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Arm O: Pralsetinib (Experimental): Participants in this treatment arm must have a positive tumor biomarker result for RET fusion.
  Interventions: Drug: Pralsetinib

INTERVENTIONS:
Drug: Entrectinib — Entrectinib will be self-administered by participants orally at home (except on clinic days), at the same time each day, on a starting dose of 600 milligrams (mg) per day once a day (QD) until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: Rozlytrek™; RG6268; RO7102122
  Arms: Arm A: Entrectinib
Drug: Inavolisib — Inavolisib will be self-administered by participants orally at home (except on clinic days) at the same time each day, on a starting dose of 9 mg/day QD until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: GDC-0077; RG6114; RO7113755
  Arms: Arm B: Inavolisib
Drug: Alectinib — Alectinib will be self-administered by participants orally at home (except on clinic days), at the same times each day, on a starting dose of 600 mg twice a day (BID) until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: Alecensa®; RG7853; RO5424802
  Arms: Arm C: Alectinib
Drug: Ipatasertib — Ipatasertib will be self-administered by participants orally at home (except on clinic days), at the same time each day, on a starting dose of 400 mg QD until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: GDC-0068; RG7440; RO5532961
  Arms: Arm D: Ipatasertib; Arm K: Ipatasertib + Atezolizumab; Arm L: Ipatasertib + Atezolizumab; Arm M: Ipatasertib + Paclitaxel
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 mg for participants on Day 1 of each 21-day cycle until unacceptable toxicity or progressive disease (or loss of clinical benefit).
  Other Names: Tecentriq®; RG7446; RO5541267
  Arms: Arm E: Atezolizumab + Investigator's Choice of Chemotherapy; Arm F: Trastuzumab Emtansine + Atezolizumab; Arm J: Trastuzumab Emtansine + Atezolizumab; Arm K: Ipatasertib + Atezolizumab; Arm L: Ipatasertib + Atezolizumab; Arm N: Atezolizumab + Tiragolumab
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered at 3.6 mg per kilogram (kg) of body weight by IV infusion every 21 days (unless dose reduction and/or dose delays are required) until disease progression or unacceptable toxicity.
  Other Names: Kadcyla®; RG3502; RO5304020
  Arms: Arm F: Trastuzumab Emtansine + Atezolizumab; Arm I: Trastuzumab Emtansine + Tucatinib; Arm J: Trastuzumab Emtansine + Atezolizumab
Drug: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf — PH FDC SC will be administered subcutaneously (SC) at a fixed non-weight-based dose. A loading dose of 1200 mg SC pertuzumab and 600 mg SC trastuzumab is then followed by a maintenance dose of 600 mg SC pertuzumab and 600 mg SC trastuzumab once every 3 weeks.
  Other Names: PHESGO™; PH FDC SC; Fixed dose combination of trastuzumab and pertuzumab administered subcutaneously; RG6264; RO7198574
  Arms: Arm G: PH FDC SC; Arm H: PH FDC SC + Investigator's Choice of Chemotherapy
Drug: Tucatinib — Tucatinib 300 mg will be administered orally BID continuously starting from Cycle 1 Day 1 onwards.
  Other Names: Tukysa™
  Arms: Arm I: Trastuzumab Emtansine + Tucatinib
Drug: Investigator's Choice of Chemotherapy — Chemotherapy will consist of docetaxel, paclitaxel, or capecitabine, as determined by the investigator, and will be administered per the respective package insert and institutional guidelines.
  Arms: Arm E: Atezolizumab + Investigator's Choice of Chemotherapy; Arm H: PH FDC SC + Investigator's Choice of Chemotherapy
Drug: Paclitaxel — The dose of paclitaxel is 80 mg/m2 administered by IV infusion on Days 1, 8, and 15 of each 28-day cycle. The paclitaxel infusion will be delivered over at least 60 minutes for each dose per institutional guidelines and administered after the oral dose of ipatasertib.
  Arms: Arm M: Ipatasertib + Paclitaxel
Drug: Tiragolumab — Following the administration of atezolizumab and an observation period, participants will receive 600 mg tiragolumab at a fixed dose administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: RG6058; RO7092284; MTIG7192A
  Arms: Arm N: Atezolizumab + Tiragolumab
Drug: Pralsetinib — Pralsetinib will be self-administered by participants orally at home (except on clinic days), at the same time each day, on a starting dose of 400 mg/day (four 100-mg capsules per day) once a day (QD) until disease progression, intolerable toxicity, or consent withdrawal.
  Other Names: GAVRETO™; RG6396; RO7499790
  Arms: Arm O: Pralsetinib

SUMMARY:
This is a Phase II, multicenter, non-randomized, open-label, multi-arm study designed to evaluate the safety and efficacy of targeted therapies as single agents or in rational, specified combinations in participants with advanced unresectable or metastatic solid tumors determined to harbor specific biomarkers.

Patients will be enrolled based on local testing performed at a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalently accredited diagnostic laboratory. The multi-arm structure of the MyTACTIC study allows patients with solid tumors to be treated with a drug or drug regimen tailored to their biomarker identified at screening.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic solid malignancy
* Positive biomarker results from a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalently accredited diagnostic laboratory and availability of a full report of the testing results. This may be from a tissue or blood sample.
* Evaluable or measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Life expectancy ≥8 weeks
* Adequate hematologic and end-organ function, as defined in the protocol, obtained within 14 days prior to initiation of study treatment
* Agrees to take measures to prevent pregnancy in the patient or partner
* In addition to the general inclusion criteria above, there are treatment-specific inclusion criteria that apply for each respective treatment arm (as detailed in the protocol)

Exclusion Criteria:

* Current participation or enrollment in another therapeutic clinical trial
* Symptomatic or actively progressing CNS metastases (asymptomatic patients with treated or untreated CNS metastases may be eligible, provided all protocol-defined criteria are met)
* History of leptomeningeal disease, unless noted otherwise for a specific treatment arm of the study
* Wide field radiotherapy within 14 days prior to start of study treatment
* Stereotactic radiosurgery within 7 days prior to start of study treatment
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infections, or any active infection that, in the opinion of the investigator, could impact patient safety
* Receipt of any anticancer drug/biologic or investigational treatment 21 days prior to Cycle 1, Day 1 except hormone therapy, which can be given up to 7 days prior to Cycle 1, Day 1 (androgen blockage may be continued for male patients with prostate cancer)
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infection with status outside of study-allowed criteria
* History of or concurrent serious medical condition or abnormality in clinical laboratory tests that precludes the patient's safe participation in and completion of the study or confounds the ability to interpret data from the study
* History of malignancy other than disease under study within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Incomplete recovery from any surgery prior to the start of study treatment that would interfere with the determination of safety or efficacy of study treatment
* Major surgical procedure, other than for diagnosis, or significant traumatic injury within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or higher), myocardial infarction, or cerebrovascular accident within 3 months prior to enrollment, unstable arrhythmias, or unstable angina
* Pregnant or breastfeeding, or intending to become pregnant during the study
* In addition to the general exclusion criteria above, there are treatment-specific exclusion criteria that apply for each respective treatment arm (as detailed in the protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (38):
- United States (38):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Arizona Clinical Research Ctr, Oro Valley, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - California Cancer Associates for Research and Excellence - Encinitas, Encinitas, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Pacific Cancer Care - Monterey, Monterey, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Kaiser Permanente Medical Ctr, Vallejo, California
  - Ventura County Hematology Oncology Specialists, Ventura, California
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Florida Cancer Specialists - PAN - SCRI - PPDS, Tallahassee, Florida
  - Florida Cancer Specialists - EAST - SCRI - PPDS, West Palm Beach, Florida
  - St Luke?s Cancer Institute, Boise, Idaho
  - Hematology and Oncology Clinic, Baton Rouge, Louisiana
  - Saint Agnes Hospital - Baltimore - Hunt - PPDS, Baltimore, Maryland
  - Ascension St. John Hospital, Detroit, Michigan
  - Frontier Cancer Center and Blood Institute, Billings, Montana
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - New Jersey Hematology Oncology Associates LLC, Brick, New Jersey
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - Central Park Hematology and Oncology, New York, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - New York Cancer & Blood Specialists, The Bronx, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Tri County Hematologyoncology, Canton, Ohio
  - SCRI Mark H. Zangmeister Center, Columbus, Ohio
  - Kaiser Permanente Center For Health Research, Portland, Oregon
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - The West Clinic, PC dba West Cancer Center, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders - PPDS, Fort Worth, Texas
  - Mays Cancer Center at UT Health San Antonio MD Anderson Cancer, San Antonio, Texas
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Northwest Medical Specialties B, Federal Way, Washington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Zuniga RM, VanderWalde A, Schwartzberg LS, Spigel DR, Passler L, Hong J, Howland M, Darbonne WC, Szado T, Daniel D. Impact of community recruitment and inclusion initiatives on enrollment in the biomarker-driven MyTACTIC trial. Future Oncol. 2026 Jan;22(1):59-69. doi: 10.1080/14796694.2025.2595690. Epub 2025 Dec 15. PMID 41392942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 252 participants with advanced unresectable or metastatic solid tumors with positive biomarker result took part in the study across 38 investigative sites in the United States.
Pre-assignment Details: Participants in this multi-arm study were treated with a drug or drug regimen tailored to their biomarker identified at screening. A total of 15 arms (Arms A to O) were planned for this study. However, no participants were enrolled in Arm A.
Groups:
- Arm B: Inavolisib (GDC-0077): Participants with a positive tumor biomarker result for phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) activating mutation self-administered inavolisib 9 milligrams (mg), orally, once a day (QD) until disease progression, intolerable toxicity, or consent withdrawal whichever occurs first.
- Arm C: Alectinib: Participants with a positive tumor biomarker result for anaplastic lymphoma kinase (ALK) gene fusion self-administered alectinib, 600 mg, orally, twice a day (BID) until disease progression, intolerable toxicity, or consent withdrawal, whichever occurs first.
- Arm D: Ipatasertib: Participants with a positive tumor biomarker result for phosphatase and tensin homolog (PTEN) loss/loss-of-function or protein kinase B (AKT) activating mutation self-administered ipatasertib, 400 mg orally, QD until disease progression, intolerable toxicity, or consent withdrawal, whichever occurs first.
- Arm E: Atezolizumab + Chemotherapy: Participants with a positive tumor biomarker result for tumor mutational burden-high (TMB-H) or microsatellite instability high (MSI-H) or deficient mismatch repair (dMMR) received atezolizumab,1200 mg, as intravenous (IV) infusion, on Day 1 of each 21-day cycle in combination with investigators choice of chemotherapy (docetaxel, paclitaxel, or capecitabine) until disease progression, loss of clinical benefit, or unacceptable toxicity whichever occurs first.
- Arm F: Trastuzumab Emtansine + Atezolizumab: Participants with a positive tumor biomarker result for human epidermal growth factor receptor 2 (HER2) gene amplification or mutation without known TMB-H/ MSI-H/ dMMR received atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle, followed by trastuzumab emtansine, 3.6 milligrams/kilograms (mg/kg), as IV infusion, every 21 days until disease progression, loss of clinical benefit, or unacceptable toxicity, whichever occurs first.
- Arm G: PH FDC SC: Participants with a positive tumor biomarker result for HER2 gene amplification or mutation without known TMB-H/ MSI-H/ dMMR received PH FDC SC, a loading dose of 1200 mg pertuzumab + 600 mg trastuzumab as subcutaneous (SC) injection on Day 1 of Cycle 1 followed by a maintenance dose of 600 mg pertuzumab + 600 mg trastuzumab as a SC injection on Day 1 of each 21-day cycle, starting at Cycle 2.
- Arm H: PH FDC SC + Chemotherapy: Participants with a positive tumor biomarker result for HER2 gene amplification or mutation without known TMB-H/ MSI-H/ dMMR received PH FDC SC, a loading dose of 1200 mg pertuzumab + 600 mg trastuzumab as a SC injection on Day 1 of Cycle 1 followed by a maintenance dose of 600 mg pertuzumab + 600 mg trastuzumab as a SC injection on Day 1 of each 21-day cycle, starting at Cycle 2 in combination with investigators choice of chemotherapy (docetaxel, paclitaxel, or capecitabine).
- Arm I: Trastuzumab Emtansine + Tucatinib: Participants with a positive tumor biomarker result for HER2 gene amplification or mutation without known TMB-H/ MSI-H/ dMMR received trastuzumab emtansine, 3.6 mg/kg as IV infusion, every 21 days in combination with tucatinib, 300 mg, orally, BID starting from Cycle 1 Day 1 until disease progression or unacceptable toxicity, whichever occurs first.
- Arm J: Trastuzumab Emtansine + Atezolizumab: Participants with a positive tumor biomarker result for HER2 gene amplification or mutation plus TMB-H/ MSI-H/ dMMR received atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle, followed by trastuzumab emtansine, 3.6 mg/kg, as IV infusion, every 21 days until disease progression, loss of clinical benefit, or unacceptable toxicity, whichever occurs first.
- Arm K: Ipatasertib + Atezolizumab: Participants with a positive tumor biomarker result for PIK3CA activating mutation received ipatasertib, 400 mg, orally QD in combination with atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit, or unacceptable toxicity, whichever occurs first.
- Arm L: Ipatasertib + Atezolizumab: Participants with a positive tumor biomarker result for PTEN loss/loss-of-function or AKT-activating mutation self-administered ipatasertib, 400 mg, orally, QD and received atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit, or intolerable toxicity, whichever occurs first.
- Arm M: Ipatasertib + Paclitaxel: Participants with a positive tumor biomarker result for co-mutations in PIK3CA activating mutations and PTEN loss/loss-of-function or AKT-activating mutation self-administered ipatasertib, 400 mg, orally, QD on Days 1 to 21 of 28-day cycles and received paclitaxel, 80 milligrams per meter square (mg/m^2), as IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, intolerable toxicity, or consent withdrawal, whichever occurs first.
- Arm N: Atezolizumab + Tiragolumab: Participants with a positive tumor biomarker result for TMB-H/ MSI-H/ dMMR received atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle, followed by tiragolumab, 600 mg, as IV infusion on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit, or unacceptable toxicity, whichever occurs first.
- Arm O: Pralsetinib: Participants with a positive tumor biomarker result for rearranged during transfection (RET) gene fusion self-administered pralsetinib, 400 mg, orally, QD until disease progression, intolerable toxicity, or consent withdrawal whichever occurs first.
Period: Overall Study
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Started | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
Completed | 2 | 3 | 5 | 4 | 5 | 4 | 0 | 5 | 3 | 4 | 5 | 1 | 6 | 1
Not Completed | 24 | 2 | 21 | 21 | 20 | 9 | 8 | 18 | 16 | 24 | 20 | 2 | 17 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 17 | 1 | 14 | 14 | 13 | 6 | 7 | 12 | 15 | 20 | 8 | 2 | 10 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Reason not Specified | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 5 | 4 | 3 | 3 | 0 | 5 | 0 | 2 | 8 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included all participants who received at least one dose of the study drug.
Groups:
- Arm B: Inavolisib (GDC-0077): Participants with a positive tumor biomarker result for PIK3CA activating mutation self-administered inavolisib 9 mg, orally, QD until disease progression, intolerable toxicity, or consent withdrawal whichever occurs first.
- Arm C: Alectinib: Participants with a positive tumor biomarker result for ALK gene fusion self-administered alectinib, 600 mg, orally, BID until disease progression, intolerable toxicity, or consent withdrawal, whichever occurs first.
- Arm E: Atezolizumab + Chemotherapy: Participants with a positive tumor biomarker result for TMB-H or MSI-H or dMMR received atezolizumab, 1200 mg, as IV infusion, on Day 1 of each 21-day cycle in combination with investigators choice of chemotherapy (docetaxel, paclitaxel, or capecitabine) until disease progression, loss of clinical benefit, or unacceptable toxicity whichever occurs first.
- Arm M: Ipatasertib + Paclitaxel: Participants with a positive tumor biomarker result for co-mutations in PIK3CA activating mutations and PTEN loss/loss-of-function or AKT-activating mutation self-administered ipatasertib, 400 mg, orally, QD on Days 1 to 21 of 28-day cycles and received paclitaxel, 80 mg/m^2, as IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, intolerable toxicity, or consent withdrawal, whichever occurs first.
- Arm O: Pralsetinib: Participants with a positive tumor biomarker result for RET gene fusion self-administered pralsetinib, 400 mg, orally, QD until disease progression, intolerable toxicity, or consent withdrawal whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib | Total
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.5) | 62.6 (6.7) | 66.7 (10.0) | 66.0 (12.0) | 66.1 (12.9) | 63.8 (10.7) | 61.1 (12.8) | 64.2 (12.0) | 61.8 (10.7) | 60.3 (10.4) | 59.8 (11.4) | 57.7 (19.4) | 63.7 (11.0) | 71.3 (16.2) | 63.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 4 | 18 | 11 | 8 | 7 | 5 | 15 | 9 | 19 | 15 | 2 | 14 | 1 | 146
  Male | 8 | 1 | 8 | 14 | 17 | 6 | 3 | 8 | 10 | 9 | 10 | 1 | 9 | 2 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 3 | 0 | 11
  Not Hispanic or Latino | 26 | 5 | 24 | 24 | 24 | 12 | 6 | 20 | 17 | 26 | 25 | 3 | 20 | 3 | 235
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 4 | 0 | 4 | 1 | 2 | 1 | 3 | 2 | 0 | 0 | 4 | 0 | 23
  White | 24 | 5 | 21 | 24 | 20 | 12 | 4 | 20 | 12 | 24 | 23 | 3 | 19 | 3 | 214
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or Response Assessment in Neuro-Oncology (RANO) Criteria for Primary Central Nervous System (CNS) Tumors
Description: Confirmed objective response rate (cORR)=percentage of participants with best response as complete response (CR) or partial response (PR) for measurable disease & CR for non-measurable disease. Confirmation=CR/PR on 2 consecutive visits ≥4 weeks apart for 3-week cycles & ≥6 weeks apart for 4-week cycles. Per RECIST, CR=disappearance of all target lesions. PR= ≥30% decrease in sum of diameters of target lesions, in absence of CR. Per RANO, CR=complete disappearance of all measurable & non-measurable disease for ≥4 weeks; no new lesions/abnormality on T2/FLAIR imaging; stable/improved non-enhancing lesions; participants must be off corticosteroids or on physiological doses; clinical status stable/improved. PR= ≥50% decrease in the sum of products of perpendicular diameters of measurable enhancing lesions on T2/FLAIR imaging for ≥4 weeks; no progression of non-measurable T1 disease; stable/improved non-enhancing lesions; corticosteroid dose ≤ baseline; clinical status stable/improved.
Time Frame: Up to 32 months
Population: Efficacy population included all participants who received at least one dose of study treatment and either had at least one post-baseline tumor assessment or discontinued treatment for any reason. Percentages have been rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
percentage of participants | 11.5 [2.4 to 30.2] | 20.0 [0.5 to 71.6] | 11.5 [2.4 to 30.2] | 28.0 [12.1 to 49.4] | 12.0 [2.5 to 31.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 36.9] | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 13.7] | 66.7 [9.4 to 99.2] | 21.7 [7.5 to 43.7] | 33.3 [0.8 to 90.6]

2. Secondary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator According to RECIST v1.1 or RANO Criteria
Description: PFS=time from start of treatment to the first occurrence of disease progression (PD) or death from any cause, whichever occurs first, per RECIST v1.1, or RANO. Per RECIST, PD=≥20% increase in sum of diameters of lesions, using the smallest sum during the study as reference, including baseline (BL). Per RANO, PD= ≥25% increase in sum of products of perpendicular diameters of enhancing lesions compared to smallest tumor measurement at BL/best response, on stable/increasing corticosteroids (CS) dose; Significant/ ≥25% increase of T2/FLAIR non-enhancing lesion on stable/increasing CS dose compared to BL/best response after therapy start; Presence of new lesions/increase of enhancement; Clear progression of non-measurable disease; Definite clinical deterioration only due to tumor/decrease in CS dose; Failure to return for evaluation due to death/deterioration. Kaplan-Meier methodology was used to estimate PFS; patients without an event were censored on the last available assessment day.
Time Frame: Time from start of treatment to the first occurrence of disease progression or death from any cause (Up to 32 months)
Population: Efficacy population included all participants who received at least one dose of study treatment and either had at least one post-baseline tumor assessment or discontinued treatment for any reason. Participants who did not experience death or disease progression were censored on the day of the last available assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
months | 4.24 [1.84 to 8.08] | 4.98 [1.54 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable because there was an insufficient number of events. | 3.48 [1.87 to 6.47] | 3.94 [2.17 to 8.38] | 4.73 [2.07 to 10.22] | 2.46 [1.77 to 5.16] | 3.02 [1.54 to 5.52] | 2.69 [1.94 to 6.18] | 1.87 [1.71 to 2.20] | 2.10 [1.64 to 3.48] | 3.61 [2.33 to 6.34] | 5.98 [1.28 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 4.76 [1.87 to 16.43] | 7.10 [1.84 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events.

3. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1 or RANO Criteria
Description: DOR was defined as the time from the date of the first confirmed complete response (CR) or partial response (PR) to disease progression (PD) or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1 or RANO. CR & PR were defined per RECIST or RANO as outlined in the description for the cORR outcome measure (OM). PD was defined per RECIST or RANO as outlined in the description for the PFS OM. Kaplan-Meier methodology was used to estimate the median DOR. The 95% confidence intervals for the median DOR were computed by the method of Brookmeyer and Crowley. Participants who did not experience death or PD were censored on the day of the last available assessment.
Time Frame: Time from the date of the first confirmed CR/PR to PD or death from any cause (Up to 32 months)
Population: Efficacy population included all participants who received at least one dose of study treatment and either had at least one post-baseline tumor assessment or discontinued treatment for any reason. Participants who achieved a confirmed CR/PR were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 3 | 1 | 3 | 7 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 5 | 1
months | 5.6 [5.3 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 6.5 [NA to NA] — The 95% CI was not estimable because only one participant had confirmed response, but the median was estimable because the participant had experienced an event. | 5.5 [3.7 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | NA [7.4 to NA] — The median and upper limit of the 95% CI was not estimable because there was an insufficient number of events. | 20.0 [NA to NA] — The 95% CI was not estimable because there was an insufficient number of events. |  |  | 7.6 [3.7 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. |  |  |  | 5.5 [4.0 to NA] — The upper limit of the 95% CI was not estimable because there was an insufficient number of events. | NA [3.6 to NA] — The median and upper limit of the 95% CI was not estimable because there was an insufficient number of events. | NA [NA to NA] — The median and 95% CI were not estimable because only one participant had confirmed response and the participant had not experienced an event (i.e., censored).

4. Secondary Outcome: PFS Rate at Month 3, 6, 9, and 12 as Determined by the Investigator According to RECIST v1.1 or RANO Criteria
Description: The PFS rates were calculated using the Kaplan-Meier (KM) method to estimate the percent survival probability of participants (i.e., PFS event-free: did not experience PD or death from any cause) in each treatment arm at landmark timepoints. The 95% confidence intervals for each PFS rate were computed by the method of Greenwood. PFS was defined as the time from the start of study treatment to the first occurrence of PD or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1 or RANO. PD was defined per RECIST or RANO as outlined in the description for the PFS OM. Participants who did not experience death or PD were censored on the day of the last available assessment. The number analyzed per landmark timepoint actually represents the number of participants who remained at risk of experiencing a PFS event at that timepoint. Percentages are rounded off to the nearest decimal point.
Time Frame: At Months 3, 6, 9 and 12
Population: Efficacy population included all participants who received at least one dose of study treatment and either had at least one post-baseline tumor assessment or discontinued treatment for any reason. The number analyzed per timepoint is the number of participants (out of the overall number of participants analyzed for PFS per arm) who remained at risk for a PFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
percent probability
  3 months: number analyzed (Participants) | 15 | 2 | 13 | 12 | 16 | 4 | 4 | 10 | 5 | 9 | 15 | 2 | 13 | 2
  3 months | 57.69 [38.7 to 76.68] | 50.00 [1.00 to 99.00] | 52.00 [32.42 to 71.58] | 52.17 [31.76 to 72.59] | 64.00 [45.18 to 82.82] | 41.03 [12.19 to 69.86] | 50.00 [15.35 to 84.65] | 48.13 [26.77 to 69.49] | 26.32 [6.52 to 46.12] | 35.56 [17.13 to 53.98] | 65.22 [45.75 to 84.68] | 66.67 [13.32 to 100.00] | 59.09 [38.55 to 79.64] | 66.67 [13.32 to 100.00]
  6 months: number analyzed (Participants) | 9 | 2 | 8 | 7 | 11 | 2 | 1 | 7 | 2 | 3 | 7 | 1 | 9 | 1
  6 months | 37.09 [18.15 to 56.03] | 50.00 [1.00 to 99.00] | 36.00 [17.18 to 54.82] | 33.20 [13.48 to 52.92] | 44.00 [24.54 to 63.46] | 20.51 [0.0 to 45.25] | 12.50 [0.00 to 35.42] | 33.69 [13.43 to 53.95] | 10.53 [0.00 to 24.33] | 11.85 [0.00 to 24.41] | 33.82 [14.13 to 53.51] | 33.33 [0.00 to 86.68] | 40.91 [20.36 to 61.45] | 66.67 [13.32 to 100.00]
  9 months: number analyzed (Participants) | 5 | 1 | 2 | 6 | 8 | 1 | 0 | 4 | 2 | 1 | 5 | 0 | 8 | 0
  9 months | 20.60 [4.61 to 36.59] | 25.00 [0.00 to 67.43] | 9.00 [0.00 to 20.78] | 28.46 [9.49 to 47.42] | 32.00 [13.71 to 50.29] | 10.26 [0.00 to 29.10] |  | 19.25 [2.32 to 36.18] | 10.53 [0.00 to 24.33] | 3.95 [0.00 to 11.53] | 24.15 [6.10 to 42.21] |  | 36.36 [16.26 to 56.46] |
  12 months: number analyzed (Participants) | 2 | 0 | 1 | 4 | 5 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 7 | 0
  12 months | 16.48 [1.79 to 31.17] |  | 4.50 [0.00 to 13.08] | 18.97 [2.39 to 35.56] | 23.33 [6.46 to 40.21] |  |  | 9.63 [0.00 to 22.30] |  |  | 14.49 [0.00 to 29.49] |  | 36.36 [16.26 to 56.46] |

5. Secondary Outcome: Percentage of Participants With Disease Control, as Determined by the Investigator According to RECIST v1.1 or RANO Criteria
Description: Disease control rate was defined as the percentage of participants whose best response was confirmed CR, confirmed PR, or a response of CR, PR, stable disease (SD), or non-CR/non-PD for a minimum of 98 days for 28-day cycle arms or 70 days for 21-day cycle arms after the first treatment date. CR & PR were defined per RECIST/RANO as outlined in the description for the cORR OM. SD per RECIST: Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. SD per RANO: Participant does not qualify for CR, PR, or minor response or PD; Stable non-enhancing (T2/FLAIR) lesions or abnormalities on same or lower dose of corticosteroids compared to baseline; No new lesions or new T2 or FLAIR abnormalities apart from those consistent with radiation effect, & no new or increased enhancement; Participants on a should be corticosteroid dose that is not greater than dose at baseline scan & is stable or improved clinically; Clinical status, stable/improved.
Time Frame: Up to 32 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
percentage of participants | 57.7 [36.9 to 76.6] | 40.0 [5.3 to 85.3] | 34.6 [17.2 to 55.7] | 32.0 [14.9 to 53.5] | 52.0 [31.3 to 72.2] | 23.1 [5.0 to 53.8] | 37.5 [8.5 to 75.5] | 26.1 [10.2 to 48.4] | 15.8 [3.4 to 39.6] | 10.7 [2.3 to 28.2] | 32.0 [14.9 to 53.5] | 66.7 [9.4 to 99.2] | 47.8 [26.8 to 69.4] | 66.7 [9.4 to 99.2]

6. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE) and Severity of AEs Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)
Description: An AE is an untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with the product. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to it. AEs were graded for severity according to NCI CTCAE v5.0. Grade 1= Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3 = Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4= Life-threatening consequences/urgent intervention indicated; Grade 5= Death related to adverse event.
Time Frame: From initiation of study drug until 28 days after the final dose of study drugs other than atezolizumab and until 90 days after the final dose of atezolizumab (Up to 32 months)
Population: Safety evaluable population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
Number analyzed (Participants) | 26 | 5 | 26 | 25 | 25 | 13 | 8 | 23 | 19 | 28 | 25 | 3 | 23 | 3
Participants
  Any Adverse Event (AE), Any Grade | 25 | 5 | 25 | 25 | 24 | 11 | 8 | 23 | 19 | 27 | 25 | 3 | 21 | 3
  Highest Severity: Grade 1 AEs | 3 | 0 | 1 | 0 | 3 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
  Highest Severity: Grade 2 AEs | 14 | 2 | 14 | 9 | 10 | 6 | 3 | 11 | 7 | 7 | 11 | 0 | 11 | 0
  Highest Severity: Grade 3 AEs | 6 | 2 | 9 | 11 | 11 | 2 | 4 | 7 | 11 | 16 | 10 | 3 | 8 | 2
  Highest Severity: Grade 4 AEs | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 0 | 0 | 0
  Highest Severity: Grade 5 AEs | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From initiation of study drug until 28 days after the final dose of study drugs other than atezolizumab and until 90 days after the final dose of atezolizumab (Up to 32 months)
Description: Safety evaluable population included all participants who received at least one dose of the study drug.
Arm/Group | Arm B: Inavolisib (GDC-0077) | Arm C: Alectinib | Arm D: Ipatasertib | Arm E: Atezolizumab + Chemotherapy | Arm F: Trastuzumab Emtansine + Atezolizumab | Arm G: PH FDC SC | Arm H: PH FDC SC + Chemotherapy | Arm I: Trastuzumab Emtansine + Tucatinib | Arm J: Trastuzumab Emtansine + Atezolizumab | Arm K: Ipatasertib + Atezolizumab | Arm L: Ipatasertib + Atezolizumab | Arm M: Ipatasertib + Paclitaxel | Arm N: Atezolizumab + Tiragolumab | Arm O: Pralsetinib
All-Cause Mortality (participants affected / at risk) | 19/26 | 1/5 | 16/26 | 16/25 | 16/25 | 6/13 | 8/8 | 14/23 | 16/19 | 22/28 | 10/25 | 2/3 | 10/23 | 1/3
Serious Adverse Events (participants affected / at risk) | 5/26 | 2/5 | 6/26 | 11/25 | 9/25 | 2/13 | 2/8 | 6/23 | 7/19 | 10/28 | 8/25 | 2/3 | 6/23 | 2/3
Other Adverse Events (participants affected / at risk) | 25/26 | 5/5 | 25/26 | 25/25 | 23/25 | 11/13 | 8/8 | 23/23 | 19/19 | 26/28 | 25/25 | 3/3 | 21/23 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B: Inavolisib (GDC-0077) (N=26) | Arm C: Alectinib (N=5) | Arm D: Ipatasertib (N=26) | Arm E: Atezolizumab + Chemotherapy (N=25) | Arm F: Trastuzumab Emtansine + Atezolizumab (N=25) | Arm G: PH FDC SC (N=13) | Arm H: PH FDC SC + Chemotherapy (N=8) | Arm I: Trastuzumab Emtansine + Tucatinib (N=23) | Arm J: Trastuzumab Emtansine + Atezolizumab (N=19) | Arm K: Ipatasertib + Atezolizumab (N=28) | Arm L: Ipatasertib + Atezolizumab (N=25) | Arm M: Ipatasertib + Paclitaxel (N=3) | Arm N: Atezolizumab + Tiragolumab (N=23) | Arm O: Pralsetinib (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B: Inavolisib (GDC-0077) (N=26) | Arm C: Alectinib (N=5) | Arm D: Ipatasertib (N=26) | Arm E: Atezolizumab + Chemotherapy (N=25) | Arm F: Trastuzumab Emtansine + Atezolizumab (N=25) | Arm G: PH FDC SC (N=13) | Arm H: PH FDC SC + Chemotherapy (N=8) | Arm I: Trastuzumab Emtansine + Tucatinib (N=23) | Arm J: Trastuzumab Emtansine + Atezolizumab (N=19) | Arm K: Ipatasertib + Atezolizumab (N=28) | Arm L: Ipatasertib + Atezolizumab (N=25) | Arm M: Ipatasertib + Paclitaxel (N=3) | Arm N: Atezolizumab + Tiragolumab (N=23) | Arm O: Pralsetinib (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (4) | 5 (7) | 5 (5) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 6 (7) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (6) | 4 (6) | 6 (6) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 7 (9) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 0 (0) | 19 (35) | 16 (20) | 3 (3) | 5 (5) | 3 (3) | 8 (13) | 3 (3) | 18 (30) | 18 (23) | 3 (7) | 4 (6) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 2 (2) | 13 (15) | 8 (10) | 6 (6) | 2 (2) | 1 (1) | 11 (15) | 6 (6) | 13 (16) | 11 (11) | 3 (5) | 10 (11) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (8) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (9) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 7 (8) | 3 (3) | 9 (10) | 6 (7) | 1 (1) | 4 (4) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 1 (1) | 5 (7) | 13 (17) | 13 (17) | 4 (4) | 1 (1) | 12 (13) | 8 (9) | 9 (11) | 12 (13) | 3 (4) | 6 (6) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 5 (5) | 0 (0) | 0 (0) | 6 (10) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 7 (9) | 0 (0) | 0 (0) | 11 (22) | 3 (3) | 1 (1) | 2 (2) | 2 (4) | 3 (4) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (6) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (4) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (5) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 6 (6) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 6 (6) | 7 (8) | 9 (11) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6) | 8 (9) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 6 (7) | 9 (10) | 2 (4) | 6 (12) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (17) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 6 (6) | 0 (0) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 5 (6) | 2 (3) | 3 (5) | 1 (1) | 0 (0) | 1 (2) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 1 (3) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (6) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (9) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 7 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 7 (9) | 4 (4) | 0 (0) | 6 (8) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin weeping (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 2 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT04632992/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04632992/SAP_001.pdf